# STUDY PROTOCOL

## 1. Study Title

Levetiracetam Versus Phenobarbitone for the Treatment of Neonatal Seizures in a Tertiary Care Hospital

Short title/acronyms: Levetiracetam Versus Phenobarbitone for the Treatment of Neonatal Seizures

#### 2. Protocol ID

DHQ-DIK-IREB NO. 4806

Date: 26 February 2024.

ClinicalTrials.gov Identifier: NCT Not Yet Assigned

## 3. Background & Rationale

Neonatal seizures are the most common neurological emergency in neonates and are associated with significant morbidity and mortality. Phenobarbitone has traditionally been the first-line anticonvulsant; however, its efficacy is limited and it has significant adverse effects. Levetiracetam is emerging as a safer alternative with promising seizure control rates. This study aims to compare the efficacy and safety of levetiracetam versus phenobarbitone in neonates with seizures.

#### 4. Objectives

#### **Primary Objective**

To compare seizure control rates within 24 hours between levetiracetam and phenobarbitone in neonates with clinically diagnosed seizures.

## **Secondary Objectives**

- To compare time to seizure cessation between both drugs.
- To compare the need for second-line anticonvulsant therapy.
- To compare seizure recurrence during hospital stay.
- To compare adverse drug reactions.
- To compare mortality rates.

#### 5. Study Design

A prospective randomized controlled trial conducted at the Neonatal Intensive Care Unit (NICU) and Pediatric wards of a tertiary care hospital.

#### 6. Study Setting

Neonatal Intensive Care Unit (NICU) and Pediatric ward at [Your Hospital Name], Pakistan.

#### 7. Study Population

Neonates (0–28 days) with clinically diagnosed seizures admitted to NICU or Pediatric ward.

### 8. Sample Size

Based on previous literature, assuming seizure control rates of 70% with levetiracetam and 50% with phenobarbitone, with 80% power and 5% significance level, the calculated sample size is  $\mathbf{n} = \mathbf{100}$  (50 in each group). However we will include all the patients accepting the inclusion criteria during one year of study.

#### 9. Inclusion Criteria

- Neonates (0–28 days old) with clinically diagnosed seizures.
- Term and preterm neonates.
- Parents/legal guardians provide informed consent.

#### 10. Exclusion Criteria

- Major congenital anomalies or genetic syndromes.
- Severe renal or hepatic impairment.
- Neonates already receiving anticonvulsants before admission.
- Neonates with metabolic seizures not responding after correction.
- Neonates with CNS infection requiring specific treatment (unless seizures persist).
- Parents refuse consent.

#### 11. Intervention

#### Arm A: Levetiracetam

- Loading dose: 20 mg/kg IV
- Repeat dose: 20 mg/kg IV after 12 hours if seizures persist
- Maintenance dose: 10 mg/kg IV/PO twice daily until seizure control or discharge

### **Arm B: Phenobarbitone**

- Loading dose: 20 mg/kg IV
- Repeat dose: 10 mg/kg IV after 20 minutes if seizures persist
- Maintenance dose: 5 mg/kg IV/PO once daily until seizure control or discharge

#### 12. Outcome Measures

# **Primary Outcome**

Seizure control rate within 24 hours after first-line treatment.

## **Secondary Outcomes**

- Time to seizure cessation
- Need for second-line anticonvulsant
- Seizure recurrence during hospital stays
- Adverse drug reactions
- Mortality during hospital stay

# 13. Study Procedures

- 1. Neonates with clinical seizures will be assessed by pediatric/neonatology team.
- 2. Eligible neonates will be randomized into either levetiracetam or phenobarbitone group.
- 3. Baseline data including demographic details, gestational age, birth weight, and clinical status will be recorded.
- 4. Standard investigations will be done (CBC, blood glucose, electrolytes, ABG, neuroimaging if required).
- 5. Treatment will be administered as per group allocation.
- 6. Monitoring of seizure activity and side effects will be done for 72 hours and until discharge.
- 7. Data will be recorded on a structured proforma.

## 14. Randomization

Simple randomization using Lottery method.

#### 15. Data Collection

Data will be collected on a structured proforma and entered into SPSS version 25.

#### 16. Ethical Considerations

Approval will be obtained from the Institutional Review Board (IRB). Informed consent will be obtained from parents/legal guardians.

# 17. Principal Investigator:

Dr. Gohar Ali